CLINICAL TRIAL: NCT06132867
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 2-Period, Crossover Study to Evaluate the Relative Bioavailability of Brigatinib Administered as an Oral Solution Versus an Immediate-Release Tablet in Adult Healthy Subjects
Brief Title: A Study to Compare the Relative Bioavailability of Brigatinib When Swallowed as a Solution Versus When Swallowed as a Tablet in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Brigatinib-1004
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): Participants received single dose of brigatinib 90 milligram (mg) as an oral solution in a fasted state on Day 1 of Period 1 (Treatment A) followed by single dose of brigatinib 90 mg as an immediate-release tablet in a fasted state on Day 1 of Period 2 (Treatment B). A washout period of at least 14 days was maintained between brigatinib administration in Period 1 and 2.
  Interventions: Drug: Brigatinib
- Sequence BA (Experimental): Participants received single dose of brigatinib 90 mg as an immediate-release tablet in a fasted state on Day 1 of Period 1 (Treatment B) followed by single dose of brigatinib 90 mg as an oral solution in a fasted state on Day 1 of Period 2 (Treatment A). A washout period of at least 14 days was maintained between brigatinib administration in Period 1 and 2.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib oral solution
Drug: Brigatinib — Brigatinib tablet
  Other Names: ALUNBRIG®

SUMMARY:
The main aim of this study is to compare the amount of brigatinib in the blood of healthy adults after they have swallowed one dose either as a solution or as a tablet.

DETAILED DESCRIPTION:
The drug being tested in this study is called brigatinib. Brigatinib is being tested to assess its relative bioavailability when administered as an oral solution versus as an immediate-release tablet in healthy participants.

The study will enroll approximately 12 participants. Participants will be randomly assigned to one of the treatment sequences:

* Sequence 1: Treatment A followed by Treatment B
* Sequence 2: Treatment B followed by Treatment A wherein Treatment A is a 90 mg oral solution dose and Treatment B is a 90 mg tablet dose.

There will be a washout period of at least 14 days between brigatinib administration in each study period. The follow-up contact will occur 14 (±2) days post the last dose of study drug.

This single-center trial will be conducted in the United States. The overall study duration is approximately 56 days.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous nonsmoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study.
2. Body mass index (BMI) ≥18.0 and ˂32.0 kilograms per meters squared (kg/m^2) at screening.
3. Pulse rate between 60 and 100 beats per minute (bpm) and a blood pressure between 90 to 140 millimeters of mercury (mmHg) systolic and 40 to 90 mmHg diastolic at screening and prior to dosing of Period 1.
4. Creatine phosphokinase is ≤1.1x upper limit of normal [ULN]; lipase, amylase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, glucose, and activated partial thromboplastin time (aPTT) are ≤ULN at screening and check-in of Period 1.

Exclusion Criteria:

1. Any history of major surgery.
2. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
3. Unable to refrain from or anticipates the use of any drug, including prescription and nonprescription medications, herbal remedies, or vitamin supplements within 28 days prior to the first dosing and throughout the study.
4. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B surface Antigen (HBsAg), or Hepatitis C Virus (HCV).
5. Positive coronavirus disease 2019 (COVID-19) results at first check-in.
6. Donation of blood or significant blood loss within 56 days prior to the first dosing.
7. Plasma donation within 7 days prior to the first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/79d6faee75ee4a31?idFilter=%5B%22Brigatinib-1004%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 20 December 2023 to 17 February 2024.
Pre-assignment Details: A total of 12 participants entered the study and were randomized in a 1:1 ratio to one of the treatment sequences: Treatment A followed by Treatment B (AB) or Treatment B followed by Treatment A (BA).
Period: Period 1 (Day 1)
Arm/Group | Sequence AB | Sequence BA
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2 (Day 1)
Arm/Group | Sequence AB | Sequence BA
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all the participants who received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence AB | Sequence BA | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (10.82) | 39.3 (8.50) | 42.3 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Brigatinib
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millliliter (ng/mL)
Groups:
- Treatment A: Brigatinib 90 mg Oral Solution: Participants received single dose of brigatinib 90 mg as an oral solution on Day 1 of Period 1 or 2 in a fasted state.
- Treatment B: Brigatinib 90 mg Tablet: Participants received single dose of brigatinib 90 mg as an immediate-release tablet on Day 1 of Period 1 or 2 in a fasted state.
Arm/Group | Treatment A: Brigatinib 90 mg Oral Solution | Treatment B: Brigatinib 90 mg Tablet
Number analyzed (Participants) | 12 | 12
nanogram per millliliter (ng/mL) | 366.6 (53.2) | 397.6 (49.7)
Statistical Analysis 1: Comparison: Treatment A: Brigatinib 90 mg Oral Solution vs Treatment B: Brigatinib 90 mg Tablet; Test type: Other — A linear mixed-effects analysis of variance model was used for the analysis. The model included sequence, treatment, and period as fixed effects and participants nested within sequence as a random effect. Geometric mean ratios and 90 percent (%) confidence intervals (CIs) were calculated using the exponentiation of the difference between treatment least square means (LSM) from the analyses on the natural log-transformed of Cmax; Geometric Mean Ratio (GMR) (%) = 92.2, 90% CI 2-sided [86.98 to 97.74] — GMR (%) was calculated as 100*(Treatment A/Treatment B)

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration for Brigatinib
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post-dose
Population: The PK analysis set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A: Brigatinib 90 mg Oral Solution | Treatment B: Brigatinib 90 mg Tablet
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*h/mL) | 6930 (43.4) | 7219 (43.6)
Statistical Analysis 1: Comparison: Treatment A: Brigatinib 90 mg Oral Solution vs Treatment B: Brigatinib 90 mg Tablet; Test type: Other — A linear mixed-effects analysis of variance model was used for the analysis. The model included sequence, treatment, and period as fixed effects and participants nested within sequence as a random effect. Geometric mean ratios and 90% CIs were calculated using the exponentiation of the difference between treatment LSM from the analyses on the natural log-transformed of AUClast; GMR (%) = 96, 90% CI 2-sided [88.48 to 104.16] — GMR (%) was calculated as 100*(Treatment A/Treatment B)

3. Primary Outcome: AUCinf: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity for Brigatinib
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Brigatinib 90 mg Oral Solution | Treatment B: Brigatinib 90 mg Tablet
Number analyzed (Participants) | 12 | 12
ng*h/mL | 7373 (39.5) | 7693 (41.0)
Statistical Analysis 1: Comparison: Treatment A: Brigatinib 90 mg Oral Solution vs Treatment B: Brigatinib 90 mg Tablet; Test type: Other — A linear mixed-effects analysis of variance model was used for the analysis. The model included sequence, treatment, and period as fixed effects and participants nested within sequence as a random effect. Geometric mean ratios and 90% CIs were calculated using the exponentiation of the difference between treatment LSM from the analyses on the natural log-transformed of AUCinf; GMR (%) = 95.84, 90% CI 2-sided [88.81 to 103.42] — GMR (%) was calculated as 100*(Treatment A/Treatment B)

4. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant who had signed informed consent form (ICF) to participate in a study. An AE can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an adverse event that was starting or worsening at the time of or after the first dose of brigatinib administered in the study. An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly or is an important medical event.
Time Frame: From first dose of the study drug up to Day 31
Population: The safety analysis set included all the participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Brigatinib 90 mg Oral Solution | Treatment B: Brigatinib 90 mg Tablet
Number analyzed (Participants) | 12 | 12
Participants
  Participants with TEAEs | 2 | 2
  Participants with SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to Day 31
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Treatment A: Brigatinib 90 mg Oral Solution | Treatment B: Brigatinib 90 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Brigatinib 90 mg Oral Solution (N=12) | Treatment B: Brigatinib 90 mg Tablet (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT06132867/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT06132867/SAP_001.pdf